CLINICAL TRIAL: NCT06318377
Title: Peanuts and Neurocognitive / Cardiovascular Health in Black Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0541
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Hypertension; Cognitive Decline; Diet; Healthy
Keywords: endothelial function; brain blood flow; cognition
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Individual will be randomly assigned either an experimental or a control condittion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peanut Consumption (Experimental): Peanuts are rich in polyphenols and also have anti-inflammatory and antioxidant properties.
  Interventions: Dietary Supplement: Peanut group
- Non-peanut consumption (No Intervention): The non-peanut consumption will simply not be consuming any additional supplements in their diet

INTERVENTIONS:
Dietary Supplement: Peanut group — These are commercially available peanuts that are high in antioxidants and are believed to be beneficial for physiological health
  Arms: Peanut Consumption

SUMMARY:
The overall research objective of this proposal is to determine the impact of increased daily peanut consumption on indices of neurocognitive and physiological health in BL individuals

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of morbidity and mortality and affects all individuals; however, its prevalence is highest in the non-Hispanic Black (BL) population. This racial disparity is present in the primary risk factors for CVD, including hypertension, atherosclerosis, and type 2 diabetes mellitus. Furthermore, this population has the highest prevalence of various neurocognitive conditions and cerebral vascular diseases including cognitive dysfunction, dementia, stroke, and Alzheimer's disease. While the association between the BL population, neurocognitive complications/cerebral vascular diseases, and CVD is multifactorial, a common link in other populations is impaired vascular function. Indeed, vascular dysfunction.

A hallmark of impaired vascular function is elevated arterial stiffness, a decrease in the vasodilator capacity, and/or heightened sympathetic vascular transduction (i.e. vasoconstrictor response and increase in peripheral vascular resistance and arterial blood pressure to efferent sympathetic neural outflow). BL individuals have impaired endothelial function evidenced by a blunted vasodilatory response to a variety of stimuli. Reduced nitric oxide (NO) bioavailability, due to elevated oxidative stress, systemic inflammation and reduced L-arginine bioavailability, is implicated as a primary contributing factor for these attenuated vasodilatory responses. Therefore, it is reasonable to speculate that an intervention targeting these pathways could abolish or minimize this elevated risk. One such intervention could be increased dietary peanut consumption which has a beneficial effect on physiological outcomes associated with neurocognitive conditions, as well as cerebral vascular and CVD risk including, cholesterol, lipid profile, insulin sensitivity / type II diabetes, cognitive health, arterial stiffness, blood pressure, and NO bioavailability and subsequently vascular function / health. However, to our knowledge the effect of increased peanut consumption on neurocognitive and CVD risk factors in the BL population remains unknown.

Therefore, the overall research objective is of this proposal is to determine the impact of increased daily peanut consumption on indices of neurocognitive and physiological health in BL individuals. The following objectives / aims will be explored:

1. Primary Aim - The primary endpoint is the effect of increased daily peanut consumption on outcomes associated with elevated risk for various neurocognitive and pathophysiological conditions/diseases. These outcomes include cognitive function, central and peripheral arterial blood pressure, cerebral and peripheral blood vessel function/health, autonomic function - i.e. vasoconstrictor responsiveness to efferent sympathetic neural outflow (sympathetic vascular transduction), and blood biomarkers (e.g., indices of inflammation, oxidative stress, insulin resistance/diabetes risk, and lipid profile).
2. Secondary Aim - A secondary endpoint is the effect of daily peanut consumption on the following variables: body composition, body weight, and body mass index (BMI).
3. Tertiary Aim - A tertiary endpoint is to examine the relationship between the various indices of physiological health with measures of Social Determinants of Health that are well known to influence the physiological outcomes that are being measured.

ELIGIBILITY:
Inclusion Criteria:

* Individuals that self-identify as white or black and who have at least one biological parent who identifies as their own self-identified race/ethnicity will be included in this study. Both men and women will be included in this study. Individuals must be between the ages of 18-50.

Exclusion Criteria:

* Individuals who have donated more than 550 ml of blood within the past 8 weeks will not have blood drawn from them in this protocol. However, if they remain interested in the study, and otherwise meet the inclusion criteria, then we may still opt to proceed with data collection.
* Individuals with peanut allergy
* Individuals in hypertensive crisis
* Pregnant women
* Breast feeding
* Allergies to spandex/lycra

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | baseline & following 8 weeks of daily peanut consumption
  Flow medicated dilation of the brachial artery
Neurocognitive Function | baseline & following 8 weeks of daily peanut consumption
  Performance on the NIH Toolbox Cognitive battery
Systolic blood pressure in brachial artery (mmHg) | baseline & following 8 weeks of daily peanut consumption
  standard blood pressure measures
Plasma concentration of total Cholesterol (Total-C) | baseline & following 8 weeks of daily peanut consumption
  assessment of total Cholesterol (Total-C)
Arterial stiffness | baseline & following 8 weeks of daily peanut consumption
  assessment of pulse wave velocity and pulse wave analysis
Diastolic blood pressure in brachial artery(mmHg) | baseline & following 8 weeks of daily peanut consumption
  standard blood pressure measures
Mean blood pressure in brachial artery (mmHg) | baseline & following 8 weeks of daily peanut consumption
  standard blood pressure measures 9(mmHg)
Plasma concentration of Low density lipoprotein (LDL) | baseline & following 8 weeks of daily peanut consumption
  assessment of Low density lipoprotein (LDL)
Plasma concentration of High density lipoprotein (HDL) | baseline & following 8 weeks of daily peanut consumption
  assessment of High density lipoprotein (HDL)
Plasma concentration of Very Low density lipoprotein (VLDL) | baseline & following 8 weeks of daily peanut consumption
  assessment of Very Low density lipoprotein (VLDL)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Brothers, PhD, Principal Investigator — University of Texas at Arlington
Locations (1):
- UT Arlington - Science and Engineering Innovation and Research Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is not plan to share IPD